CLINICAL TRIAL: NCT07085429
Title: Development of a Prospective Monocentric Clinico-Biological Database for Bronchial Cancer
Brief Title: Development of Clinical and Biological Database on Bronchial Cancer
Acronym: BCBPoumon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2021-11 BPO
Record Dates: First submitted 2025-07-02; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Bronchial Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Bronchogenic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchial cancer (Experimental): Additionnal samples from routine care of different natures (blood, tumor tissue ans healthy tissue) and standardized clinical data will be entered into a database.
  Interventions: Biological: Blood and tissue sampling

INTERVENTIONS:
Biological: Blood and tissue sampling — Tissue samples (tumor tissue and healthy tissue) frozen and secured in paraffin collected during surgery.
  During the blood samples taken for diagnosis and / or treatment when possible. Additional samples for research purposes will be carried out, these blood samples will be collected:
  * before any therapeutic intervention (T1) for a total volume of 36mL,
  * prior to surgery (T-Surg) for a total volume of 24mL,
  * at each progression (T2a, b, c…) for a total volume of 24mL,
  * at the end of follow-up (T3) for a total volume of 24mL.

SUMMARY:
A Clinical and Biological Database will provide to the scientific community a collection of blood and tissues with clinical data to improve knowledge about cancer and help to develope new cancer treatments. This database is specific to bronchial cancer.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related mortality and the third most commonly diagnosed cancer. In France in 2018, it accounted for 46,363 new cases and 33,117 deaths. The overall 5-year survival rate across all stages and sexes is 20%.

Diagnosis is most often made at the metastatic stage, which significantly worsens the prognosis. Since 2020, the standard treatment for such cases has been the administration of intravenous chemo-immunotherapy, in the absence of a molecular alteration that allows for access to an oral targeted therapy. Immunotherapy and targeted therapies have considerably improved the prognosis for some patients, but the vast majority experience therapeutic resistance, either early or delayed.

The prognostic and predictive mechanisms of treatment response are poorly understood and vary greatly between histological and molecular subtypes. It is therefore crucial to gain a better understanding of these mechanisms in order to ultimately identify new therapeutic avenues to improve patient outcomes.

The first step in this process is to establish a tissue and blood biobank from patients with bronchial carcinoma (both small-cell and non-small-cell) treated at our center.

The Clinical Biological DataBase (BCB) is a tool:

* for research in analytical and public health epidemiology, biological research and for the development of data useful for clinical research and therapeutic trials;
* to help scientists understand and explain phenomena ranging from the interaction of molecules to the whole metabolism of the organism in normal and pathological situations;
* to identify potential strategies for prevention, diagnosis, management and analysis of cancer subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged over 18 years,
* Histologically or cytologically confirmed bronchial cancer,
* Treatment-naïve patient for the current cancer,
* Patient who has provided informed, written, and explicit consent,
* Patient affiliated with the French national health insurance system.

Exclusion Criteria:

* Patient with a WHO performance status ≥ 3,
* Pregnant and/or breastfeeding woman,
* Patient with a history of other cancers within the 5 years preceding inclusion,
* Patient for whom regular follow-up is considered impossible due to psychological, familial, social, or geographic reasons,
* Patient under legal protection (guardianship, curatorship, or judicial protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who consent to participate in the study | through study completion : an average of 1 year
  the proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France, France